CLINICAL TRIAL: NCT02777515
Title: Pilot Study of the Immediate Cardiovascular Effects of Electronic Cigarette in Subjects With Cardiovascular Disease
Brief Title: Study of the Immediate Cardiovascular Effects of Electronic Cigarette in Subjects With Cardiovascular Disease
Acronym: ECLOPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ECLOPE
Record Dates: First submitted 2016-05-09; First posted 2016-05-19 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: CARDIOVASCULAR DISEASES
Keywords: electronic cigarette
MeSH Terms: conditions — Cardiovascular Diseases; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients using electronic cigarette (Other): The patients under the age of 35 followed at the consultation of rythmology for a cardiovascular assessment and already smoking the electronic cigarette and this since at least 1 month. The patient will receive a clinical examination, an electrocardiogram, a Holter-ECG and an echocardiogram before and after electronic cigarette consumption for 15 minutes.
  Interventions: Behavioral: using electronic cigarette

INTERVENTIONS:
Behavioral: using electronic cigarette — Assesment of patients, using electronic cigarette, presenting to the Rhythm of consultation for a cardiovascular evaluation by:
  1. A compendium of history, a general physical examination (weight, height) and cardiovascular with measurement of oxygen saturation, an assessment of past and current smoking (with documentation of the concentration of nicotine in the electronic cigarette and the product brand used)
  2. measurement of blood pressure
  3. An electrocardiogram
  4. A Holter-ECG 10 minutes
  5. A transthoracic echocardiogram

SUMMARY:
Justification Smoking is a major factor for mortality and cardiovascular morbidity. The electronic cigarette, sometimes presented as smoking cessation "classic" is expanding but its safety has not been established to date. The smoke from the electronic cigarette is mainly composed of propylene glycol, some adverse effects were observed in animals.

Study Type interventional study assessing the effect of the electronic cigarette Inclusion criteria Topics under 35 years presenting to Rhythm of the consultation for a cardiovascular evaluation and already smoking the electronic cigarette and that for at least 1 month

Exclusion criteria

* Consumption of traditional cigarettes, nicotine replacement or toxic
* Presence of heart disease Primary objective To evaluate in a pilot study the immediate cardiovascular effects of electronic cigarette consumption Number of patients 20 Duration of Study Recruitment in 2015 for an unlimited period of inclusion. Exam time is about two hours.

Procedures performed during the study Physical examination, ECG, Holter-ECG 10 minutes and echocardiography were performed before and 15 minutes after the consumption of the usual electronic cigarette of the subject.

No additional follow-up visit is required

DETAILED DESCRIPTION:
I. Introduction

The objective of this study was to evaluate the acute cardiovascular effects of electronic cigarette in young patients by non-invasive methods.

II. State of the question and justification for the research

State of the question

Coronary artery disease is the death rate cause, responsible for around 7 million deaths each year, or 12.8% of causes of death. Myocardial infarction has an incidence of 66/100 000 inhabitants per year. It is now undoubtedly recognized that smoking is a major independent cardiovascular risk factor and tobacco is responsible for over 5 million deaths per year.

Inhaled tobacco is harmful because it contains several components: nicotine, tar derivatives, derived free radicals nitric oxide and carbon monoxide. The acute effects of smoking on the cardiovascular system are complex. The effects on the coronary circulation are characterized by decreased blood flow intracoronary, particularly in patients with underlying coronary artery disease, exacerbating myocardial ischemia. There is also a detrimental effect on systolic and diastolic function of the left ventricle, from the first flashes. Tobacco alters peripheral resistance and promotes the secretion of adrenergic catecholamines.

Smoking cessation is naturally a public health priority but remains difficult because of the addictive nature of nicotine. Thus several substitutes for the cessation assistance were developed, among them the electronic cigarette is a recent option, more and more fashionable.

Study Rationale

The safety of the electronic cigarette is not established yet. There are only rare small number of studies comparing mostly acute cardiovascular effects of electronic cigarette to those of the conventional cigarette without analyzing all the potential consequences of the electronic cigarette.

The smoke from the electronic cigarette is mainly composed of propylene glycol, also with nicotine in varying concentrations. Propylene glycol is used as a filling liquid of electronic cigarettes and is usually considered harmless if inhaled, despite having been cause asystole, shock and decreased renal and pulmonary arterial flow after intravenous injection in calves. It is also used by the food industry as an emulsifier or as a solvent for certain liquid aromas. Its cardiovascular effects are clearly not been studied in humans.

The interest of our study was to evaluate the acute cardiovascular effects of electronic cigarette, with simple, non-invasive means.

III. population concerned

Defined in th eligibility section.

IV. Study Methodology

Recruitment is expected from H1 2015. Patients will be recruited during the Heart Rhythm consultation for a cardiovascular evaluation. We plan to include a minimum of 20 subjects. After this first phase of recruitment, data analysis will be conducted to determine if there instead of increasing the number of subjects to be included.

A cardiovascular evaluation will be conducted at baseline, including:

1. A compendium of history, a general physical examination (weight, height) and cardiovascular with measurement of oxygen saturation, an assessment of past and current smoking (with documentation of the concentration of nicotine in the electronic cigarette and the product brand used)
2. measurement of blood pressure
3. An electrocardiogram (ECG)
4. A Holter-ECG 10 minutes
5. A transthoracic echocardiogram

   The ECG will analyze heart rate, time of conduction and repolarization (QT interval in particular).

   The Holter ECG will study the heart rate variability in a short time.

   Echocardiography (15) will assess o cardiac output: measurement of sub aortic Integral time speed ITS o diastolic function of the left ventricle: measurement of peak E wave 'and the wave in tissue Doppler to the mitral annulus; mitral profile measurement with the peak of the E wave, the deceleration time, the peak of the A wave and the E / A ratio; measuring the peaks of the S wave and D, pulmonary S / D ratio

   o end-systolic and end-diastolic volume of the left ventricle with assessment of systolic left ventricular function (LVEF)
   * systolic function of the right ventricle: the measurement wave S tricuspid annulus and tricuspid annular plane systolic excursion (TAPSE) section 4 cavities, measuring SPSP

   A recent study showed that a significant level of nicotine in the blood was reached after 10 puffs right from the 10th minute after the first puff. This rate is then growing for one hour, when the inhalation continues. For practical reasons, we will ask the subjects to smoke for 15 minutes at their usual pace.

   Cardiac evaluations described above will be repeated. The duration of this review is about two hours.

   To minimize bias, ECG, Holter-ECG and echocardiography will be stored anonymously and interpreted retrospectively by a physician blinded to the patient's identity and time of completion (before or after inhalation) for each examination.

   V. Data Privacy

   Written information will be given about. Her signed consent will be collected and stored.

   For each subject an identifier will be given for exams before inhalation and another identifier will be given for the examinations after inhalation. These identifiers will be graded on a handwritten sheet without data entry.

   The anonymous data will then be entered on a computer file which will be sent to the statistician in charge of the analysis. There will be no exchange of personal data.

   VI. Statistical analysis

   Quantitative variables are expressed by their mean, standard deviations, their minimum and maximum values as appropriate. The variables will be expressed in numbers and percentages.

   The purpose of statistical analysis will determine if there is a significant difference of the variables collected from pre and post-inhalation inhalation of cigarette smoke electronic period.

   VII. Vigilance

   at. definitions

i. adverse Event

Any untoward medical occurrence that occurs in a person who is ready to biomedical research that this event is related or not to research or (x) product (s) on the (s) is (s) door this research.

ii. Serious Adverse Event (SAE)

A serious event is an event:

* The evolution of which is fatal; or
* Which endangers the life of the person undergoing research; or
* Which causes a disability or a significant or lasting disability; or
* Causing hospitalization or prolongation of hospitalization; or
* Which results in an abnormality or birth defect; or
* Any other event does not meet the qualifications listed above, but can be regarded as "potentially serious" including some laboratory abnormalities; or
* Medically relevant event in the judgment of the investigator; or
* Events requiring medical intervention to prevent progression to one of the aforementioned states.

The term "life-threatening" is reserved for immediate life-threatening at the time of the adverse event, regardless of the consequences of corrective or palliative therapy.

Certain circumstances requiring hospitalization are not within the gravity standard "inpatient / hospitalization extension" as:

admission for social or administrative reasons; hospitalization predefined by the protocol; hospitalization for medical or surgical treatment scheduled prior research; passing day hospital.

b. detection methods and collection of adverse events

All adverse events should be investigated, reported and recorded, processed and evaluated the first visit (inclusion D0) until the end of the study until their resolution. Adverse events are collected:

* In clinical, biological and other planned and systematic examination by the investigator;
* By spontaneous reporting by the participants, who will be instructed to contact the investigating doctor in case of adverse events.

All adverse events will be recorded on forms on adverse events of case report form (see Appendix 2). Each observed adverse events will be recorded individually. The intensity of adverse events will be determined as follows:

* Mild (grade 1): no interference on the daily activity of the patient;
* Moderate (grade 2): Moderate interference on the patient's daily activities but still acceptable;
* Severe (grade 3) significant interference on the patient's daily activity and unacceptable;
* Threat of life-threatening (grade 4);
* Death (Grade 5). All adverse events must be graded. Responsibilities of the investigator.

  i. Declaration of SAEs

The investigator evaluates each adverse event in relation to its severity. The investigator must notify by fax (01 44 12 31 40) to the sponsor (CRC GHPSJ) without delay after the day he heard, all serious adverse events in the trial, except from those identified in the protocol as not requiring immediate reporting. This initial notification is the subject of a written report must be followed if necessary by one or the report (s) Additional (s) writing (s) Main (s) within 8 days of the first declaration (Declaration Form in Annex 3 of the Protocol).

The investigator must document the best event (thanks to copies of laboratory results or reports of examinations or hospitalization accounts informing the serious event, including relevant negative results, not forgetting to make these documents and anonymous to register number and the patient's code), medical diagnosis and a causal link between serious adverse events and research.

The statement is sent to the developer with the serious adverse event reporting form signed and dated.

The investigator should follow the patient with an SAE to its resolution, stabilization at a level deemed acceptable by the investigator or return to the previous state, even if the patient is out of the test and inform the promoter (CRC GHPSJ) by fax on 01 44 31 December 40 with the form (check: monitoring).

ii. Assessment of causality

The investigator should assess causality of adverse events with research. The causal link is binary (connected / not connected).

iii. Reporting period and followed the terms of adverse events

The investigator should report serious adverse events from the inclusion of the patient until the end of the experimental procedure.

The investigator should monitor adverse events until resolution or stabilization even if the patient is out of the study.

iv. Special cases

2.4.1 Serious Events not immediately declare To the extent it is expected no serious adverse event related to the participation of patients in this study and that only certain serious adverse events known to be associated with the patient's usual care may arise, these will therefore not require immediate declaration in accordance with the health authorities.

c. Responsibilities promoter

The Promoter will declare to ANSM (French Health Authorities) and the CPP (patients protection committee) in accordance with the law of 9 August 2004:

• all unexpected serious adverse reactions without delay and at the latest within seven calendar days from the day when the sponsor becomes aware of, and within 7 days for monitoring,

* developments without delay safety and at the latest within 7 calendar days, and within 7 days for monitoring,
* annual safety reports within 60 calendar days of the anniversary date of the study.

  d. Establishment of an independent oversight committee

To the extent it is expected no serious adverse event related to the participation of patients in this study, we do not want to establish an independent monitoring committee.

VIII. Funding

No external funding GHPSJ.

IX. Conflicts of interest

No conflict of interest

ELIGIBILITY:
Inclusion Criteria:

* Aged under 35 years
* Having no known heart disease
* Not consuming any toxic
* Already smoking the electronic cigarette and that for at least one month to ensure good tolerance of the electronic cigarette

Exclusion Criteria:

* Subjects also smoking a conventional cigarette or using other nicotine substitutes will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2015-12-05 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of change of blood pressure | before smoking then 15 min after smoking
Assessment of change of Electrocardiogram (ECG) | before smoking then 15 min after smoking
Assessment of change of Holter-ECG | before smoking then 15 min after smoking
Assessment of change of transthoracic echocardiogram | before smoking then 15 min after smoking

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan MOUBARAK, MD, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France